CLINICAL TRIAL: NCT01873014
Title: the Effect of Chinese Herbs to Treat Thyroid Diseases With Different Iodine Intake
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: head2012neck
Record Dates: First submitted 2013-03-07; First posted 2013-06-07 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2012-05

CONDITIONS: Thyroid Diseases
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high Iodine intake (Experimental)
  Interventions: Drug: chinese herbs-I
- low Iodine intake (Active Comparator)
  Interventions: Drug: chinese herbs-II

INTERVENTIONS:
Drug: chinese herbs-I — two agent per day, twice a day
  Arms: high Iodine intake
Drug: chinese herbs-II — two agent per day, twice a day
  Arms: low Iodine intake

SUMMARY:
safe study of Chinese Herbs to Treat Thyroid Diseases With Different Iodine

DETAILED DESCRIPTION:
Based on the previous studies, the research choose the patients with different iodine intake,and improve our original Chinese Herbs thyroid III formula, in order to provide the patients the best individual treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* patient with thyroid diseases

Exclusion Criteria:

* not meet the diagnostic criteria,women with pregnancy or lactation ,drug allergy ,need surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
diameter，number of the tumor | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: yu yang, doctor, Study Director — doctor